CLINICAL TRIAL: NCT04736459
Title: Does Pre-washing the Catheter With a Culture Medium Before Intrauterine Insemination Have an Effect on Pregnancy Rates?
Brief Title: Pre-washing the Catheter With a Culture Medium Before Intrauterine Insemination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Vehbi Yavuz Tokgoz, Assocciate Professor, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2222392979
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Infertility
Keywords: intrauterine insemination, pre-washing catheter
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Washed Catheter (Experimental): Washed catheter arm: will be washed with culture medium before insemination
  Interventions: Procedure: Pre-washed catheter vs. Unwashed catheter in the intrauterine insemination
- Unwashed Catheter (Sham Comparator): Unwashed catheter arm: will not be washed with culture medium.
  Interventions: Procedure: Pre-washed catheter vs. Unwashed catheter in the intrauterine insemination

INTERVENTIONS:
Procedure: Pre-washed catheter vs. Unwashed catheter in the intrauterine insemination — The pre-washed catheter will be washed with culture medium before intrauterine insemination The unwashed catheter will not be washed with culture medium as a standard intrauterine insemination procedure

SUMMARY:
The aim of the study to evaluate the possible effect of washing the insemination catheters before intrauterine insemination on the pregnancy outcomes.

We know that washing the catheters are already washed in the case of embryo transfer for assisted reproductive techniques. Based on this knowledge, we also constituted the hypothesis which is about the impact of washing the catheter on the gametes and embryos. The pre-washing the catheter before intrauterine insemination may provide higher pregnancy results.

ELIGIBILITY:
Inclusion Criteria:

* at least 1-year infertility
* at least one patent fallopian tube confirmed by hysterosalpingography (HSG) or laparoscopy
* ovulatory menstrual cycles
* suitable semen analysis according to the World Health Organization (WHO) criteria for intrauterine insemination

Exclusion Criteria:

* bilateral tubal occlusion
* mild or severe endometriosis
* day 3 serum FSH (follicle-stimulating hormone) > 13 IU/L
* abnormal thyroid function tests, hyperprolactinemia
* total motile sperm count (TMSC) < 5 millions or severe teratospermia (<4% normal forms) following semen preparation
* more than 3 follicles above the size of 17mm on the day of ovulation triggering

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-29 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 8 weeks after intrauterine insemination
  Clinical pregnancy will be defined as the presence of a heartbeat at 6th gestational weeks

IPD SHARING:
Plan to Share IPD: No